CLINICAL TRIAL: NCT02112292
Title: The Role of the Endocannabinoid System in Sweet Taste Intensity and Liking
Acronym: Sweed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL44758.081.13; 2013-002555-14 (EudraCT Number)
Record Dates: First submitted 2014-03-25; First posted 2014-04-11 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Sensory Science
MeSH Terms: interventions — Dronabinol; Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- T-C-P (Experimental): Order of administrations: tetrahydrocannabinol - cannabidiol - placebo
  Interventions: Drug: tetrahydrocannabinol; Drug: cannabidiol; Drug: Placebo
- T-P-C (Experimental): Order of administrations: tetrahydrocannabinol - placebo - cannabidiol
  Interventions: Drug: tetrahydrocannabinol; Drug: cannabidiol; Drug: Placebo
- C - T - P (Experimental): Order of administrations: cannabidiol - tetrahydrocannabinol - placebo
  Interventions: Drug: tetrahydrocannabinol; Drug: cannabidiol; Drug: Placebo
- C - P - T (Experimental): Order of administrations: cannabidiol - placebo - tetrahydrocannabinol
  Interventions: Drug: tetrahydrocannabinol; Drug: cannabidiol; Drug: Placebo
- P - T - C (Experimental): Order of administrations: placebo - tetrahydrocannabinol - cannabidiol
  Interventions: Drug: tetrahydrocannabinol; Drug: cannabidiol; Drug: Placebo
- P - C - T (Experimental): Order of administrations: placebo - cannabidiol - tetrahydrocannabinol
  Interventions: Drug: tetrahydrocannabinol; Drug: cannabidiol; Drug: Placebo

INTERVENTIONS:
Drug: tetrahydrocannabinol
  Other Names: delta-9-tetrahydrocannabinol; THC
Drug: cannabidiol
  Other Names: CBD
Drug: Placebo

SUMMARY:
The endocannabinoid (eCB) system, a neurochemical signalling system consisting of CB-receptors and their endogenous ligands, has been found to be involved in food intake of sweet and palatable foods. Activation of the eCB system increases food intake and vice versa. The mechanism behind this effect is still unknown and the current study aims at clarifying why sweet food intake increases. It is hypothesized that sweet taste intensity increases and that sweet taste is experienced as more pleasant.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 18.5 - 25 kg/m2
* Incidental cannabis use for at least one year, at least four times per year, but less than once a week.
* Dutch-speaking
* Willing to comply with the study procedures
* Having given written informed consent

Exclusion Criteria:

* Not meeting the inclusion criteria
* Restraint eating (men: score > 2.90)
* Lack of appetite
* Having difficulties with swallowing/eating
* Usage of an energy restricted diet during the last two months
* Weight loss or weight gain of 5kg or more during the last two months
* Stomach or bowel disease
* Diabetes, thyroid disease, other endocrine disorders
* Use of daily medication except paracetamol
* Having taste or smell disorders (self-report)
* Being allergic/intolerant for products under study
* Previously experienced an adverse reaction to cannabinoids (e.g. anxiety, paranoia, nausea)
* Having (had) a schizophrenia or other psychotic illness
* Having a family history of schizophrenia or other psychotic illness
* Working at the Division of Human Nutrition (WUR)
* Current participation in other research from the Division of Human Nutrition (WUR)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04-16 (Actual); Study Completion 2015-04-16 (Actual)

PRIMARY OUTCOMES:
Relation between sweet taste intensity and liking | 15 minutes after intervention
  The main study parameter is the relation between sucrose intensity scaling (psychophysics) and liking (psychohedonics) of drinks with the different sucrose concentrations. These scores will be assessed after six participants and at end of the study.

SECONDARY OUTCOMES:
Ranking order of pleasantness of different drinks with different levels of sucrose. | 25 minutes after intervention
  Ranking order will be assessed after 6 participants and at end of the study
Preferences for different kinds of foods | 45 minutes after intervention (15 minutes after top-up dose)
  Preference for foods high in one of three macronutrients (carbohydrate, protein, fat) or low in energy
Ad libitum intake | 35 minutes after intervention (5 minutes after top-up dose)
  Ad libitum intake of a chocolate-based drink
Change of plasma levels of (endo-)cannabinoids and satiety hormones | One hour after intervention
Polymorphisms | At test session, i.e., 2 weeks before first intervention
  The genetic determination of the enzymes responsible for the metabolism of THC and CBD.

OTHER OUTCOMES:
Descriptives | At inclusion of participants
  General subject characteristics, e.g age, restrained eating score and other lifestyle and medical parameters
Appetite ratings | During each test session
  During each test session, appetite ratings will be assessed at several time points
Subjective feelings | During each test session
  During each test sessions, participants will rate the effects of the intervention.
Perception | 20 minutes after intervention
  Participants will rate the intensity of different shades of grey.
Sweet taste intensity | 15 minutes after intervention
  Sucrose intensity of drinks (psychophysics) of drinks with different sucrose concentrations. This will be assessed after six participants and at end of the study.
Liking of sweet taste | 15 minutes after intervention
  Liking (psychohedonics) of drinks with the different sucrose concentrations. This will be assessed after six participants and at end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne EM de Bruijn, MSc, Principal Investigator — Wageningen University; Gerry Jager, Dr., Study Chair — Wageningen University
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands